CLINICAL TRIAL: NCT06375343
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of PRO-240 Ophthalmic Solution Compared to Optive® on the Ocular Surface of Ophthalmologically and Clinically Healthy Volunteers
Brief Title: Study to Evaluating PRO-240 Ophthalmic Solution Compared to Optive®
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOPH240-0923/I
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease; Dry Eye Sensation; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, comparative, single-blind, single-center, comparative clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-240 (Experimental): * Propylene glycol 0.3% - Polyethylene glycol 400 0.5% - Glycerin 0.2%. Ophthalmic solution.
  * Dosage: 1 drop QID [4] (four times per day) for 7 days in both eyes.
  * Route of administration: Ophthalmic
  Interventions: Drug: PRO-240
- Optive® (Active Comparator): * Carboxymethylcellulose 0.5%; Glycerin 0.9%. Ophthalmic solution.
  * Dosage: 1 drop QID [4] (four times per day) for 7 days in both eyes.
  * Route of administration: Ophthalmic
  Interventions: Drug: Optive®

INTERVENTIONS:
Drug: PRO-240 — -Propylene glycol 0.3%, Polyethylene glycol 400 0.5%, and Glycerin 0.2%. Ophthalmic solution.
  Arms: PRO-240
Drug: Optive® — - Carboxymethylcellulose 0.5%, and Glycerin 0.9%. Ophthalmic solution.
  Arms: Optive®

SUMMARY:
This is a phase I clinical study to evaluating safety and tolerability of PRO-240 ophthalmic solution through the incidence of unexpected adverse events, as well as through changes in Best Corrected Visual Acuity (BCVA), and the incidence of stinging after its administration, compared to Optive®.

DETAILED DESCRIPTION:
The variables to be evaluated include:

Primary (safety):

- Incidence of unexpected advere events (AE's)

Secondary:

* Changes in the ocular comfort index (OCI) score
* Changes in intraocular pressure (IOP)
* Changes in Best Corrected Visual Acuity (BCVA)
* Adherence to treatment
* Changes in tear film breakup time
* Changes in fluorescein staining
* Changes in lissamine green staining

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Ophthalmologically and clinically healthy subjects.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age ≥18 years.
* Male or female gender.
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the informed consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Best corrected visual acuity (BCVA) of 20/30 or better in both eyes.
* Corneal staining ≤ grade I on the Oxford Scale.
* Having an intraocular pressure ≥ 10 and ≤ 21 mmHg.

Exclusion Criteria:

* History of hypersensitivity to any of the components of the drugs under investigation.
* Use of ophthalmic medications from any pharmacological group.
* Use of medications by any other route of administration.
* Use of non-steroidal anti-inflammatory drugs, steroid anti-inflammatory drugs, or antibiotics by any route of administration in the last 30 days.
* History of eye surgery in the last 6 months.
* Use of contact lenses for a period less than two weeks prior to the start of the study, and during the intervention period of this study.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* History of any chronic-degenerative disease, including Diabetes Mellitus or Systemic Arterial Hypertension.
* Diagnosis of glaucoma or ocular hypertension.
* Known diagnosis of liver or heart disease.
* Presenting active inflammatory or infectious disease at the time of entry into the study.
* Presenting unresolved lesions or traumas at the time of entry into the study.
* Having been subjected to non-ophthalmological surgical procedures in the last 3 months.
* Being or having an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an employee of the research site or the sponsor, and who directly participates in this study.
* Active smoking (specified as the consumption of cigarettes regardless of the amount and frequency, 4 weeks prior to study inclusion and during the intervention period of this study).
* Active alcoholism (specified as the consumption of alcoholic beverages, regardless of the amount and frequency, 72 hours prior to study inclusion and during the intervention period of this study).

Elimination Criteria:

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of unexpected adverse events related to the interventions | Days 0: (Basal Visit), 8 (Final Visit) and 11 (Safety Call)
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.

SECONDARY OUTCOMES:
Changes in the Ocular Comfort Index score | Days: 0 (Basal Visit), and 8 (Final Visit)
  Changes in the Ocular Comfort Index (OCI) score in between interventions, the subjects will be questioned regarding this symptoms' incidence. The OCI contains 8 items (one positive and eight negative) that focus on discomfort associated with ocular surface disorders. Each of these questions has two parts, which separately inquire about the frequency and severity of symptoms.
  The OCI score will be used for evaluation of tolerability through incidence and severity of dry eye symptoms in a scale from 0 to 100. Greater scores mean a worse outcome.
Adherence to treatment (adherence) Adherence to treatment (adherence) | Days: 8 (Final Visit)
  Adherence will be evaluated through the treatment record in the subject's diary.
Changes in Best Corrected Visual Acuity (BCVA) | Days: 0 (Basal Visit) and 8 (Final Visit)
  The BCVA will be evaluated through Snellen chart.
Changes in tear film breakup time | Days: 0 (Basal Visit) and 8 (Final Visit)
  The most common method for assessing stability is with fluorescein. The precorneal layer colored with fluorescein will change to less fluorescent or non-fluorescent regions. The time from the last blink to the appearance of these regions is the tear film breakup time.
Changes in intraocular pressure (IOP) | Days: 0 (Basal Visit) and 8 (Final Visit)
  Previous instillation of topical anesthetic, the IOP will be measured through a Goldmann tonometer during visits
Changes in the integrity of the ocular surface (fluorescein staining) | Days: 0 (Basal Visit) and 8 (Final Visit)
  Changes in the integrity of the ocular surface using fluorescein staining and evaluated through the Oxford scale. The standard Oxford scale for fluorescein staining has the following criteria: Grade 0- Equal to or less than panel A; Grade I- Equal to or less than panel B, greater than panel A; Grade II- Equal to or less than panel C, greater than panel B; Grade III- Equal or less than panel D, greater than panel C; Grade IV- Equal or less than panel E, greater than panel D; Grade V- Greater than panel E.
Changes in lissamine green staining of the conjunctival surface | Days: 0 (Basal Visit) and 8 (Final Visit)
  Direct observation with slit lamp, graded according to (changes in ocular surface staining using the Sjögren's International Collaborative Clinical Alliance [SICCA].)

IPD SHARING:
Plan to Share IPD: No